CLINICAL TRIAL: NCT04872244
Title: Results of Intrauterine Levonorgestrel Use for the Patients With Isthmocele Suffering From Postmenstrual Spotting Without Fertility Desire
Brief Title: Can Intrauterine Levonorgestrel Releasing Device Be a Treatment Option for Postmenstrual Spotting in Isthmocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma ketenci gencer, Dr., Gaziosmanpasa Research and Education Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GaziosmanpasaTREHB
Record Dates: First submitted 2020-06-15; First posted 2021-05-04 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-06

CONDITIONS: Isthmocele; Post-menstrual Spotting Bleeding; Pelvic Pain
Keywords: isthmocele; postmenstrual spotting bleeding; pelvic pain
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Intervention Model Description: patients who have isthmocele due to previous cesarean section and suffering from postmenstrual spotting bleeding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- patients with isthmosele that mirena ( levonorgestrel releasing intrauterine device) was applied (Experimental): outcome measures of patients suffering from postmenstruel spotting due to ısthmosele whom mirena ( levonorgestrel releasing intrauterine device) was applied
  Interventions: Device: usage of mirena ( levonorgestrel releasing intrauterine device) in isthmocele; Drug: Levonorgestrel Drug Implant Product

INTERVENTIONS:
Device: usage of mirena ( levonorgestrel releasing intrauterine device) in isthmocele — usage of mirena ( levonorgestrel releasing intrauterine device) in isthmocele for postmenstrual spotting and do not have desire for fertility
  Other Names: levonorgestrel
Drug: Levonorgestrel Drug Implant Product — intrauterine administration

SUMMARY:
it was planned to investigate the treatment effect of levonorgestrel releasing intrauterine device in patient with isthmocele who were suffering from postmenstrual spotting bleeding and who had no desire for fertility.

DETAILED DESCRIPTION:
isthmocele is an acquired diverticulum like defect of myometrium in the anterior isthmic part of uterus due to previous cesarean section incision. It can be defined as thinning of the incised site of uterus smaller than 50 % of its normal thickness. the real incidence is unknown. due to low ability of contractility of the postmenstrual spotting bleeding. Accumulation of blood in the isthmocele induces inflammation within the endometrium and causes pain as well. Furthermore, this inflammation can be an absolute reason for secondary infertility. As a result, accumulation of blood in the isthmocele seems to start up the cascade of morbidities. When understanding the mechanism, preventing blood accumulation seems to prevent symptoms other than infertility. Levonorgestrel releasing intrauterine devices can be a way of thinning the endometrium hence, blood accumulation can be avoided. In the literature, surgical correction of the isthmocele has been studied and medical treatment that was mentioned in the literature was the oral contraceptives and only a preliminary report of very small sample size, discussed the effect of levonorgestrel releasing device . in the light of aforementioned clinical knowledge, we planned to investigate the treatment effect of levonorgestrel releasing intrauterine device in patients with postmenstrual bleeding due to isthmocele who were not willing to have baby. These patients will be called back at 6th, 12th and 18th months after applying levonorgestrel releasing device to the uterus. Gynecological examinations will be done and complainants will be questioned.

ELIGIBILITY:
Inclusion Criteria:

* having isthmocele and complaining for postmestrual spotting bleeding
* having cesarean section as a last delivery way.
* not planning for fertility
* complaining about dysmenorrhea and pelvic pain

Exclusion Criteria:

* having pelvic infection
* having an any type of previous pelvic surgery
* having leiomyoma, endometrial polyp or adnexal mass
* having any type of malignancy
* having thyroid dysfunction and prolactinemia

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
incidence of postmenstrual spotting bleeding | 18 months
  incidence of vaginal spotting bleeding after normal menstrual bleeding
incidence of dysmenorrhea | 18 months
  incidence of pelvic pain felt by the patient during mensturation
incidence of pelvic pain | 18 months
  incidence of pelvic pain regardless of mensturation

CONTACTS AND LOCATIONS:
Locations (1):
- saglik Bilimleri Univercity Gaziosmanpaşa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided